CLINICAL TRIAL: NCT00000671
Title: A Phase II Efficacy Study Comparing 2',3'-Dideoxyinosine (ddI) (BMY-40900) and Zidovudine Therapy of Patients With HIV Infection Who Have Been on Long Term Zidovudine Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Bristol-Myers Squibb (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: ACTG 117; 070V1; AI454-009
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2011-03-14 (Estimated); Status verified 1992-08

CONDITIONS: HIV Infections
Keywords: Didanosine; Zidovudine
MeSH Terms: conditions — HIV Infections | interventions — Zidovudine; Didanosine

INTERVENTIONS:
Drug: Zidovudine
Drug: Didanosine

SUMMARY:
To compare the effectiveness and toxicity of didanosine (ddI) and zidovudine (AZT) in patients with AIDS or advanced AIDS-related complex (ARC) who have tolerated AZT therapy for 12 months or longer. Per amendment, asymptomatic patients with CD4 counts less than 200 cells/mm3 are eligible.

AZT is effective in reducing mortality in patients with AIDS who receive the drug after the first episode of Pneumocystis carinii pneumonia (PCP) and in patients with advanced ARC. However, AZT therapy has been associated with significant toxicities. In addition, the effectiveness of AZT appears to decrease during the second and third years of therapy. For these reasons, the development of alternative therapy that would be at least as effective but less toxic is of great importance. The drug ddI is an antiviral agent that inhibits replication of HIV with less apparent toxicity than AZT. Studies indicate that ddI remains active in the body for at least 12 hours; thus benefits of ddI might be achieved with a low frequency of drug administration.

DETAILED DESCRIPTION:
AZT is effective in reducing mortality in patients with AIDS who receive the drug after the first episode of Pneumocystis carinii pneumonia (PCP) and in patients with advanced ARC. However, AZT therapy has been associated with significant toxicities. In addition, the effectiveness of AZT appears to decrease during the second and third years of therapy. For these reasons, the development of alternative therapy that would be at least as effective but less toxic is of great importance. The drug ddI is an antiviral agent that inhibits replication of HIV with less apparent toxicity than AZT. Studies indicate that ddI remains active in the body for at least 12 hours; thus benefits of ddI might be achieved with a low frequency of drug administration.

Two dose levels of ddI, each adjusted depending on patient's weight at study entry, are compared with a variable dosage regimen of AZT (the dose which the patient is tolerating at the time of study entry). Randomization is stratified by baseline CD4 cell count (less than 100 or 100-300) and Medical Center. This study continues for at least 12 months after the entry of the first subject. Patients randomized to AZT will receive orally. All patients randomized to AZT also receive a ddI placebo at 12 hour intervals. Patients randomized to ddI receive AZT placebo.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Required:

* Aerosolized pentamidine (300 mg every 4 weeks).

Allowed:

* Chronic suppressive treatment for toxoplasmosis, Pneumocystis carinii pneumonia (PCP), cryptococcal meningitis, herpes simplex virus infection.
* Ganciclovir for patients developing cytomegalovirus (CMV) infection while in study.
* Erythropoietin for patients under the relevant treatment IND.
* Treatment of opportunistic infections with other than sulfonamide-containing regimens.
* Aspirin, acetaminophen, or non-steroidal anti-inflammatory agents is discouraged, but is permitted for as short a period of time as possible.
* Chronic use of trimethoprim - sulfamethoxazole or other sulfonamide preparations is not encouraged while on study.

Patients must:

* Have had the diagnosis of AIDS or advanced AIDS related complex (ARC).
* Have received AZT therapy for at least 12 months, with a minimal daily dose of 500 mg/day and with no more than 60 days off AZT therapy within the 12 month period; medical records with documentation of AZT dosing must be provided.
* Provide informed consent (guardian as appropriate).
* Be available for follow-up for at least 6 months.
* Have the inclusion laboratory values within approximately 14 days of initiating therapy (except for CD4 cell counts).
* Patients whose AIDS-defining condition is Kaposi's sarcoma alone must have CD4 cell counts < 300 cells/mm3.

Allowed:

* Positive blood culture for Mycobacterium avium or Cytomegalovirus.
* Prior history of toxoplasmosis, Herpes simplex, Cryptococcus, or Pneumocystis carinii pneumonia (PCP) requiring chronic suppressive therapy.
* Occasional premature atrial or ventricular contractions.

Prior Medication:

Required:

* Zidovudine (AZT) therapy for at least 12 months, with a minimal daily dose of 500 mg/day, and with no more than 60 days off AZT therapy within the 12-month period (documentation of AZT dosing must be provided).

Allowed:

* Intralesional agents.

Exclusion Criteria

Co-existing Condition:

Patients with the following are excluded:

* Psychological or emotional problems sufficient, in the investigator's opinion, to prevent adequate compliance with study therapy.
* AIDS-dementia complex = or > stage 2.
* Active AIDS defining opportunistic infections not specifically allowed.
* Intractable diarrhea.
* Grade 2 neuropathy, based on the Neuropathy Targeted Symptom Questionnaire, or any moderate abnormality indicative of peripheral neuropathy, particularly impaired sensation of sharp pain, light touch, or vibration in the lower extremities, distal extremity weakness, or distal extremity hyperreflexia.
* Prior history of acute pancreatitis within past 2 years or chronic pancreatitis.
* History of seizures within past 2 years or currently requiring anticonvulsants for control.
* History of past or current heart disease.
* Malignancy likely in the investigator's opinion to require cytotoxic chemotherapy during the expected course of this trial.
* Life expectancy < 3 months.

Concurrent Medication:

Excluded:

* Isoniazid (INH). Neurotoxic drugs. Oral acidifying agents.

Patients with the following are excluded:

* Psychological or emotional problems sufficient, in the investigator's opinion, to prevent adequate compliance with study therapy.
* AIDS-dementia complex = or > stage 2.
* Active AIDS defining opportunistic infections not specifically allowed.
* Intractable diarrhea.
* Prior history of acute pancreatitis within past 2 years or chronic pancreatitis.
* History of seizures within past 2 years or currently requiring anticonvulsants for control.
* History of past or current heart disease.
* Malignancy likely in the investigator's opinion to require cytotoxic chemotherapy during the expected course of this trial.
* Life expectancy = or < 3 months.
* Previous participation in any study of ddI, ddC or d4T.

Prior Medication:

Excluded:

* Ganciclovir (DHPG).
* Excluded within 1 month of study entry:
* ddI and any other antiretroviral drug or investigational anti-HIV agent except for zidovudine (AZT).

Interferons.

* Immunomodulating drugs.
* Cytotoxic agents not specifically allowed.
* Neurotoxic drugs.

Excluded within 3 months of study entry:

* Ribavirin.

Prior Treatment:

Excluded within 14 days of study randomization:

* Blood transfusion.

Active alcohol or drug abuse that is sufficient, in investigator's opinion, to prevent adequate compliance with study therapy.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 750
Dates: Primary Completion 1992-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J Kahn, Study Chair; D Richman, Study Chair
Locations (71):
- United States (70):
  - Children's Hosp of Los Angeles/UCLA Med Ctr, Los Angeles, California
  - Los Angeles County - USC Med Ctr, Los Angeles, California
  - Cedars Sinai / UCLA Med Ctr, Los Angeles, California
  - UCLA CARE Ctr, Los Angeles, California
  - Harbor - UCLA Med Ctr / UCLA School of Medicine, Los Angeles, California
  - Palo Alto Veterans Adm Med Ctr / Stanford Univ, Palo Alto, California
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - San Francisco AIDS Clinic / San Francisco Gen Hosp, San Francisco, California
  - Stanford at Kaiser / Kaiser Permanente Med Ctr, San Francisco, California
  - Stanford Univ School of Medicine, Stanford, California
  - Olive View Med Ctr, Sylmar, California
  - Sepulveda Veterans Adm Med Ctr / Olive View Med Ctr, Sylmar, California
  - Harbor UCLA Med Ctr, Torrance, California
  - Mountain States Regional Hemophilia Ctr / Univ of Colorado, Denver, Colorado
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - George Washington Univ Med Ctr, Washington D.C., District of Columbia
  - G E Morey Jr, Fort Lauderdale, Florida
  - Univ of Miami School of Medicine, Miami, Florida
  - Northwestern Univ Med School, Chicago, Illinois
  - Rush Presbyterian - Saint Luke's Med Ctr, Chicago, Illinois
  - Edward Hines Veterans Administration Hosp, Hines, Illinois
  - Indiana Univ Hosp, Indianapolis, Indiana
  - Univ of Kansas School of Medicine, Wichita, Kansas
  - Louisiana Comprehensive Hemophilia Care Ctr, New Orleans, Louisiana
  - Louisiana State Univ Med Ctr / Tulane Med School, New Orleans, Louisiana
  - Tulane Univ School of Medicine, New Orleans, Louisiana
  - Harvard (Massachusetts Gen Hosp), Boston, Massachusetts
  - Boston Med Ctr, Boston, Massachusetts
  - Beth Israel Deaconess - West Campus, Boston, Massachusetts
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Baystate Med Ctr of Springfield, Springfield, Massachusetts
  - Med Ctr of Central Massachusetts, Worcester, Massachusetts
  - Univ of Massachusetts Med Ctr, Worcester, Massachusetts
  - Univ of Minnesota, Minneapolis, Minnesota
  - Nebraska Regional Hemophilia Ctr, Omaha, Nebraska
  - SUNY / Erie County Med Ctr at Buffalo, Buffalo, New York
  - City Hosp Ctr at Elmhurst / Mount Sinai Hosp, Elmhurst, New York
  - Beth Israel Med Ctr / Peter Krueger Clinic, New York, New York
  - Bellevue Hosp / New York Univ Med Ctr, New York, New York
  - Cornell Univ Med Ctr, New York, New York
  - Mem Sloan - Kettering Cancer Ctr, New York, New York
  - Saint Luke's - Roosevelt Hosp Ctr, New York, New York
  - Mount Sinai Hemophilia Ctr / Mount Sinai Med Ctr, New York, New York
  - Mount Sinai Med Ctr, New York, New York
  - Univ of Rochester Medical Center, Rochester, New York
  - SUNY - Stony Brook, Stony Brook, New York
  - SUNY / State Univ of New York, Syracuse, New York
  - Bronx Municipal Hosp Ctr/Jacobi Med Ctr, The Bronx, New York
  - Jack Weiler Hosp / Bronx Municipal Hosp, The Bronx, New York
  - Montefiore Med Ctr / Bronx Municipal Hosp, The Bronx, New York
  - Bronx Veterans Administration / Mount Sinai Hosp, The Bronx, New York
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Duke Univ Med Ctr, Durham, North Carolina
  - Bowman Gray School of Medicine / Wake Forest Univ, Winston-Salem, North Carolina
  - Holmes Hosp / Univ of Cincinnati Med Ctr, Cincinnati, Ohio
  - Univ Hosp of Cleveland / Case Western Reserve Univ, Cleveland, Ohio
  - Ohio State Univ Hosp Clinic, Columbus, Ohio
  - Med College of Ohio, Toledo, Ohio
  - Milton S Hershey Med Ctr, Hershey, Pennsylvania
  - Univ of Pennsylvania, Philadelphia, Pennsylvania
  - Hemophilia Ctr of Western PA / Univ of Pittsburgh, Pittsburgh, Pennsylvania
  - Univ of Pittsburgh Med School, Pittsburgh, Pennsylvania
  - Julio Arroyo, West Columbia, South Carolina
  - Univ of Tennessee / E Tennessee Comprehensive Hemophilia Ctr, Knoxville, Tennessee
  - Hermann Hosp / Univ Texas Health Science Ctr, Houston, Texas
  - Dr Stephen L Green, Hampton, Virginia
  - Univ of Washington, Seattle, Washington
  - Dr Brian Buggy, Milwaukee, Wisconsin
  - Milwaukee County Med Complex, Milwaukee, Wisconsin
  - Great Lakes Hemophilia Foundation, Milwaukee, Wisconsin
- San Juan Veterans Administration Med Ctr, San Juan, Puerto Rico

REFERENCES:
- [Background] Smith MS, Koerber KL, Pagano JS. Long-term persistence of zidovudine resistance mutations in plasma isolates of human immunodeficiency virus type 1 of dideoxyinosine-treated patients removed from zidovudine therapy. J Infect Dis. 1994 Jan;169(1):184-8. doi: 10.1093/infdis/169.1.184. PMID 7506280
- [Background] Bozzette SA, Hays RD, Berry SH, Kanouse DE. A Perceived Health Index for use in persons with advanced HIV disease: derivation, reliability, and validity. Med Care. 1994 Jul;32(7):716-31. doi: 10.1097/00005650-199407000-00005. PMID 8028406
- [Background] Fiscus SA, Heggem-Snow A, Troiani L, Wallmark E, Folds JD, Sheff B, van der Horst CM. Transient high titers of HIV-1 in plasma and progression of disease. J Acquir Immune Defic Syndr Hum Retrovirol. 1995 May 1;9(1):51-7. PMID 7712235
- [Background] Coombs RW, Welles SL, Hooper C, Reichelderfer PS, D'Aquila RT, Japour AJ, Johnson VA, Kuritzkes DR, Richman DD, Kwok S, Todd J, Jackson JB, DeGruttola V, Crumpacker CS, Kahn J. Association of plasma human immunodeficiency virus type 1 RNA level with risk of clinical progression in patients with advanced infection. AIDS Clinical Trials Group (ACTG) 116B/117 Study Team. ACTG Virology Committee Resistance and HIV-1 RNA Working Groups. J Infect Dis. 1996 Oct;174(4):704-12. doi: 10.1093/infdis/174.4.704. PMID 8843206
- [Background] Richardson D, Liou SH, Kahn JO. Uric acid and didanosine compliance in AIDS clinical trials: an analysis of AIDS Clinical Trials Group protocols 116A and 116B/117. J Acquir Immune Defic Syndr (1988). 1993 Nov;6(11):1212-23. PMID 8229656
- [Background] Kozal M, Winters M, Shafer R, Kroodsma K, Katzenstein D, Merigan T. Behavior of codon 74 and 215 pol gene mutations in 62 AZT experienced patients on ddI monotherapy. Natl Conf Hum Retroviruses Relat Infect (1st). 1993 Dec 12-16;55
- [Background] Kozal MJ, Kroodsma K, Winters MA, Shafer RW, Efron B, Katzenstein DA, Merigan TC. Didanosine resistance in HIV-infected patients switched from zidovudine to didanosine monotherapy. Ann Intern Med. 1994 Aug 15;121(4):263-8. doi: 10.7326/0003-4819-121-4-199408150-00005. PMID 7518658
- [Background] Schooley RT. Correlation between viral load measurements and outcome in clinical trials of antiviral drugs. AIDS. 1995 Dec;9 Suppl 2:S15-S19. PMID 8775802
- [Background] Kahn JO, Lagakos SW, Richman DD, Cross A, Pettinelli C, Liou SH, Brown M, Volberding PA, Crumpacker CS, Beall G, et al. A controlled trial comparing continued zidovudine with didanosine in human immunodeficiency virus infection. The NIAID AIDS Clinical Trials Group. N Engl J Med. 1992 Aug 27;327(9):581-7. doi: 10.1056/NEJM199208273270901. PMID 1353607
- [Background] Richman DD. Clinical significance of drug resistance in human immunodeficiency virus. Clin Infect Dis. 1995 Oct;21 Suppl 2:S166-9. doi: 10.1093/clinids/21.supplement_2.s166. PMID 8845446